CLINICAL TRIAL: NCT04897516
Title: Phase III Randomized,Multicenter Non-inferiority Study to Evaluate the Efficacy and Safety of Shorter Benznidazole Regimens Compared to the Standard Regimen to Treat Adult Patients With Chronic Chagas Disease
Brief Title: Shorter Benznidazole Regimens Compared to the Standard Regimen for Chagas Disease
Acronym: NuestroBen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NuestroBen
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-09

CONDITIONS: Chagas Disease
Keywords: Chagas disease; Benznidazole; Trypanosoma Cruzi; Standar treatment; Short treatment
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Intervention Model Description: Phase III, open-label, prospective, controlled, multicenter, non-inferiority study to compare the efficacy of the Drug: 1. Short regimen of benznidazole :Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 2 weeks.
  2. Drug: Short regimen of benznidazole : Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 4 weeks. And 3. Drug: Standard treatment with benznidazole : Benznidazole, 300 mg divided into three daily doses (100 mg every 08 hours), orally for 8 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Short regimen of benznidazole 2 weeks (Experimental): Experimental: Short regimen of benznidazole Participants will receive an investigational treatment of benznidazole for 2 weeks.
  Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 2 weeks.
  Interventions: Drug: Short regimen of benznidazole
- Short regimen of benznidazole 4 weeks (Experimental): Experimental: Short regimen of benznidazole Participants will receive an investigational treatment of benznidazole for 4 weeks.
  Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 4 weeks.
  Interventions: Drug: Short treatment with benznidazole
- Standard treatment with benznidazole (Active Comparator): Active Comparator: Standard treatment with benznidazole Benznidazole, 300 mg divided into three daily doses (100 mg every 08 hours), orally for 8 weeks
  Interventions: Drug: Standard treatment with benznidazole

INTERVENTIONS:
Drug: Short regimen of benznidazole — Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 2 weeks.
  Other Names: Benznidazole 2 weeks
  Arms: Short regimen of benznidazole 2 weeks
Drug: Short treatment with benznidazole — Benznidazole, under the brand name Abarax (100 mg tablet), 300 mg divided into three daily doses (100 mg every 08 hours) for 4 weeks.
  Other Names: Benznidazole 4 weeks
  Arms: Short regimen of benznidazole 4 weeks
Drug: Standard treatment with benznidazole — Benznidazole, 300 mg divided into three daily doses (100 mg every 08 hours), orally for 8 weeks
  Other Names: Benznidazole 8 weeks
  Arms: Standard treatment with benznidazole

SUMMARY:
Chagas disease, a parasitic infection caused by Trypanosoma cruzi, is endemic in much of Latin America and affects people throughout the world. Currently treatment with the only two drugs effective against the infection, benznidazole and nifurtimox, has significant limitations including frequent adverse effects in adult patients. However, timely treatment is key to achieving global objectives of controlling the disease. The standard treatment has a long duration (60 days). NuestroBen will test the hypothesis that shorter treatment regimens of 14 days and 28 days will be non-inferior to the standard 60-day treatment while improving the safety profile.

DETAILED DESCRIPTION:
Chagas disease is a vector-borne parasitic infection affecting an estimated 6 million people worldwide. Very few people have been able to access antiparasitic treatment for the disease, and about 20% of those who do initiate treatment are unable to complete it due to the long duration (2 months) and side effects associated with the current regimen. Benznidazole is one of only two drugs with proven efficacy against Trypanosoma cruzi, the parasite that causes the disease. An earlier Phase 2 clinical trial, BENDITA, indicated 89% of 30 patients treated with a shorter (2-week) regimen of benznidazole maintained sustained parasite clearance after 12 months of follow-up, with no discontinuations of treatment due to side effects. The current study will evaluate shorter treatment regimens with benznidazole in a Phase III clinical trial. NuestroBen will assess the efficacy and safety of 2-week and 4-week regimens of BZN (300 mg daily), compared to the standard treatment of BZN 300 mg daily for 8 weeks, in terms of reducing and eliminating the T. cruzi parasite in adults in the chronic phase of Chagas disease with the indeterminate form or mild cardiac progression. Efficacy will be measured through conversion from positive to negative parasitaemia according to the results of qualitative PCR tests from the end of treatment, and up to 12 months of follow-up from the end of treatment. Safety will be compared according to the frequency and severity of adverse events. Patients adherence to treatment in each study arm will also be described.

ELIGIBILITY:
Inclusion criteria (Subjects must meet ALL the inclusion requirements listed below to enter the study):

* Signed informed consent form;
* Between ≥18 and ≤60 years of age;
* Weight ≥ 50 kg to ≤ 95 kg;
* Confirmation of the diagnosis of T. cruzi infection by conventional serology (a minimum of two tests must be reactive);
* Serial qualitative PCR (one blood sample divided in three DNA extractions, at least one of which must be positive);
* Women of childbearing potential must have a negative pregnancy result at the time of inclusion, must not be breast-feeding, and must use a highly effective method of contraception during study treatment and until 30 days after the last dose of study treatment or demonstrate permanent sterilization;
* Ability to comply with all exams and specific protocol visits;
* Having a permanent address;
* ECG criteria: (Heart rate: 50 -100 bpm or isolate sinus bradycardia from 41 to 59 beats/min; QRS ≤120 msec, and QTc ≥ 350 msec and ≤ 450 msec) at screening) or following findings belonging to non-severe chagasic cardiomyopathy: uncomplete right bundle branch block, Left anterior fascicular block, First-degree atrioventricular block, Low voltage. The abnormalities included are not exclusionary;
* Normal or minimal structural changes in echocardiogram (left ventricular diastolic diameter (LVDD) <= 55 mm, diastolic dysfunction, absence of Microaneurysm or tip aneurysm, absence of hypo or generalized akinesia, absence of Systolic dysfunction (low fractional shortening and ejection fraction), and/or absence of mural thrombus);
* Not presenting signs or symptoms of moderate- severe chronic cardiac and/or digestive forms of Chagas disease (criteria detailed in Study Manual and specific SOP);
* No prior history of mental disorders or suicidal tendencies;
* Not suffering from known acute or chronic illnesses at the moment of selection for the study that, in the Investigator's discretion, may interfere with the evaluation of the efficacy or safety of the investigational product (such as acute infections, immunosuppressive conditions, or liver or kidney diseases that have required treatment);
* Not having received a formal indication not to take BZN (contraindication, according to the Summary of Product Characteristics - SmPC);
* No prior history of hypersensitivity, allergy, or serious adverse reactions to any of the nitroimidazole compounds (including BNZ) and/or its components/excipients;
* Have not previously undergone antiparasitic treatment for T. cruzi infection;
* No prior history of drug abuse or alcoholism;
* Not suffering from any disease or condition that prevents subjects from consuming oral medication.

Exclusion criteria (The presence of any of the items below will exclude subjects from inclusion in the study):

* Subject pregnant or intending to become pregnant during treatment and within 30 days of the last dose of study treatment;
* Signs or symptoms of the established (moderate- severe) chronic cardiac and/or digestive form of Chagas disease, or any ECG/ echocardiographic findings not included at Inclusion criteria;
* History of cardiomyopathy, heart failure, or severe ventricular arrhythmia;
* History of digestive surgery potentially related to Chagas Disease or megacolon / mega-esophagus;
* Acute or chronic disease that, in the Investigator's discretion, may interfere with the evaluation of the efficacy or safety of the investigational product (such as acute infection, history of immunosuppressive conditions, or liver or kidney disease that has required treatment);
* Laboratory test values that are considered clinically significant or outside the allowable values, per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1;
* Disease or clinical condition that prevents subjects from consuming oral medication;
* Subjects with a contraindication (known hypersensitivity) to any of the nitroimidazole compounds, e.g. metronidazole;
* Subjects with a history of allergy (serious or not), allergic rash, asthma, intolerance, sensitivity or photosensitivity;
* Concomitant use and/or consumption of allopurinol, antimicrobial and antiparasitic agents, herbal medicines, dietary supplements and energy drinks;
* Scheduled surgery that may interfere with the conduct of the trial and/or with the treatment evaluation;
* Inability to attend study visits, comply with treatment, and cooperate with study procedures;
* Previous participation in a trial for the evaluation of the treatment of T. cruzi infection;
* Simultaneous participation in another trial or within 3 months prior to screening for this trial (in accordance with national regulations).
* Subjects suffering from a serious medical or psychiatric illness that increases the risk associated with study participation or that interferes with the interpretation of study results should not be included.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with sustained negativation of parasitemia according to the results of qualitative PCR tests | From the end of treatment, and up to 12 months of follow-up from the end of treatment.
  Sustained parasitological response will be determined by negative serial qualitative PCR results (two negative PCR results from three DNA extractions from a sample) from the end of treatment with the elimination of sustained parasitaemia until the end of 12 months' follow-up from the end of treatment.

SECONDARY OUTCOMES:
Proportion of patients with negative parasitemia at 1, 4, 6 and 8 months follow-up form the end of treatment | 1, 4, 6 and 8 months from the end of treatment
  Proportion of patients with negative parasitemia at 1, 4, 6 and 8 months follow-up form the end of treatment
Incidence and severity of adverse events | From the end of treatment, and up to 12 months of follow-up from the end of treatment
  Incidence and severity of adverse events
Incidence of SAEs, Adverse Events of Special Interest (AESIs) and/or adverse events that cause treatment interruption | From the end of treatment, and up to 12 months of follow-up from the end of treatment.
  Incidence of SAEs, Adverse Events of Special Interest (AESIs) and/or adverse events that cause treatment interruption
Descriptions of patients adherence to treatment in each study arm. | 2, 4 and 8 weeks
  describing the number of completed treatment in patients vs uncompleted treatment in patients

OTHER OUTCOMES:
Incidence and severity of adverse events | From the end of treatment, and up to 12 months of follow-up from the end of treatment.
  Incidence and severity of adverse events
Incidence of SAEs, Adverse Events of Special Interest (AESIs) and/or adverse events that cause treatment interruption | From the end of treatment, and up to 12 months of follow-up from the end of treatment
  Incidence of SAEs, Adverse Events of Special Interest (AESIs) and/or adverse events that cause treatment interruption

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Pinazo, MD, Study Director — Drugs for Neglected Diseases
Locations (6):
- Argentina (6):
  - Instituto Nacional de Parasitología "Dr. Mario Fatala Chaben", Buenos Aires
  - Fundación Huésped, Buenos Aires
  - Hospital Francisco Javier Muñiz, Buenos Aires
  - Hospital Donación Francisco Santojanni, Buenos Aires
  - Instituto de Cardiología de Corrientes "Juana Francisca Cabral", Corrientes
  - Centro de Chagas y Patología Regional, Hospital Independencia, Santiago del Estero

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be made available upon request. Requests are evaluated by DNDi's scientific advisory committee. Interested researchers can contact DNDi for data access requests via email at ctdata@dndi.org. Researchers can also request data by completing the form available at https://www.dndi.org/category/clinical-trials/. In this data request form, researchers must confirm that they will share data and results with DNDi and will publish any results open access.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of study results
Access Criteria: Beginning 6 months after publication of study results

REFERENCES:
- [Derived] Marques T, Forsyth C, Barreira F, Lombas C, Blum de Oliveira B, Laserna M, Molina I, Bangher MDC, Javier Fernandez R, Lloveras S, Fernandez ML, Scapellato P, Patterson P, Garcia W, Ortiz L, Schijman A, Moreira OC, Garcia L, Viele K, Longhi S, Vaillant M, Tipple C, Fraisse L, Silvestre-Sousa A, Sosa-Estani S, Pinazo MJ. New regimens of benznidazole for the treatment of chronic Chagas disease in adult participants in indeterminate form or with mild cardiac progression (NuestroBen study): protocol for a phase III randomised, multicentre non-inferiority clinical trial. BMJ Open. 2025 Sep 30;15(9):e098079. doi: 10.1136/bmjopen-2024-098079. PMID 41027700